For Protocol Amendment #03 to: NRG-GY027

NCI Protocol #: NRG-GY027 Local Protocol #: NRG-GY027 NCI Version Date: 12/22/2023

## SUMMARY OF CHANGES

| # | Section | Comments |
|---|---|---|
| 1 | Title Pages | NCI Version Date is now 12/22/2023 |
| 2 | [What are the | This section has been updated to note the end of the escalation phase |
| | study | and the opening of the dose expansion phase after having determined |
| | groups?] | the MTD. |

# **Research Study Informed Consent Document**

**Study Title for Participants:** Testing the addition of a new drug Ipatasertib to the usual chemotherapy treatment (paclitaxel and carboplatin) for ovarian cancer.

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: PROTOCOL NRG-GY027, "PHASE I/IB SAFETY AND PHARMACODYNAMIC STUDY OF NEOADJUVANT (NACT) PACLITAXEL AND CARBOPLATIN WITH IPATASERTIB AS INITIAL THERAPY OF OVARIAN CANCER PTMA 100805" (NCT# 05276973)

## **Overview and Key Information**

## What am I being asked to do?

We are asking you to take part in a research study. This study has public funding from the National Cancer Institute (NCI), part of the National Institutes of Health (NIH) in the United States Department of Health and Human Services. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

We are asking you to take part in this research study because you have newly diagnosed epithelial ovarian cancer.

## Taking part in this study is your choice.

You can choose to take part or you can choose not to take part in this study. You also can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document has important information to help you make your choice. Take time to read it. Talk to your doctor, family, or friends about the risks and benefits of taking part in the study. It's important that you have as much information as you need and that all your questions are answered. See the "Where can I get more information?" section for resources for more clinical trials and general cancer information.

# Why is this study being done?

This study is being done to answer the following question:

Can we improve the treatment outcomes of your ovarian cancer by adding ipatasertib to the usual combination of chemotherapies (paclitaxel and carboplatin)?

We are doing this study because we want to test the safety of a drug called ipatasertib at different doses.

- 1 -

Protocol Version Date: 12/22/2023

# What is the usual approach to my ovarian cancer?

The usual approach for patients who are not in a study is your physician's choice of treatment using the FDA approved drugs paclitaxel and carboplatin.

## What are my choices if I decide not to take part in this study?

- You may choose to have the usual approach described above.
- You may choose to take part in a different research study, if one is available.
- You may choose not to be treated for cancer.
- You may choose to only get comfort care to help relieve your symptoms and not get treated for your cancer.

## What will happen if I decide to take part in this study?

If you decide to take part in this study, a sample of your tumor that was removed during a previous surgery or biopsy will be submitted. Then you will take the study drug ipatasertib by mouth every day in addition to usual chemotherapy (paclitaxel and carboplatin) of treatment. Then you will continue to take ipatasertib alone for an additional before having surgery to remove the ovarian tissue, a procedure that is the usual standard of care. A portion of your tumor will also be used for testing.

After you finish your treatment, your doctor and study team will watch you for side effects at clinic visits or by phone if you are unable to visit the clinic. These follow up visits will occur 30 days after the last day of treatment and again 90 days after the last day of treatment. If there are any side effects that lead to discontinuing the treatment, then you will be followed until you recover.

# What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important for you to think carefully about these as you make your decision.

#### **Risks**

We want to make sure you know about a few key risks right now. We give you more information in the "What risks can I expect from taking part in this study?" section.

If you choose to take part in this study, there is a risk that the addition of ipatasertib may not be as good as the usual approach at preventing your cancer from growing or coming back.

There is also a risk that you could have side effects from the study drug ipatasertib. These side effects may be worse and may be different than you would get with the usual approach for


cancer. There is a risk in delay of standard of care debulking surgery if serious AEs occur due to combination of investigational ipatasertib with neoadjuvant therapy.

Some of the most common side effects that the study doctors know about are:

- Allergic reaction
- Diarrhea
- Vomiting, Nausea
- Fatigue
- Sores in the mouth which may cause difficulty swallowing
- Loss of appetite

There may be some risks that the study doctors do not yet know about.

#### **Benefits**

There is some evidence in people with other types of cancer that adding ipatasertib to the usual approach can lower the chance of your tumor growing or spreading for longer than the usual approach alone. However, we do not know if this will happen in people with ovarian cancer. We do not know if adding ipatasertib to the usual approach will help you live longer than the usual approach alone. This study may help the study doctors learn things that may help other people in the future.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop taking part in the study at any time.

If you decide to stop, let your study doctor know as soon as possible. It's important that you stop safely. This may mean slowly stopping the study drugs so that there is not a sudden unsafe change or risk to your health. If you stop, you can decide if you want to keep letting the study doctor know how you are doing.

There are two options of stopping treatment:

- 1. The first option is that you stop treatment, but you would continue follow up visits (no treatment) to see how you are doing. If you agree to let your study doctor continue to follow you, you will continue to be part of the study so that we can follow you to see how you are doing and if your cancer comes back. We would continue to collect information about how you and your cancer are doing and to see how the treatment affected you and your cancer. This is considered that you go "off treatment" but not "off study" and you would not withdraw consent.
- 2. The second option is to stop treatment and not allow your study doctor to collect any information on how you and your cancer are doing and how the treatment affected you and your cancer. This is considered "withdrawal of consent" and you would go "off treatment" and "off study".

- 3 -


Your study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes and the study is no longer in your best interest.
- New information becomes available and the study is no longer in your best interest.
- You do not follow the study rules.
- You become pregnant while on the study.
- The study is stopped by the Institutional Review Board (IRB), Food and Drug Administration (FDA), or study sponsor NCI (National Cancer Institute). The study sponsor is the organization who oversees the study.

It is important that you understand the information in the informed consent before making your decision. Please read, or have someone read to you, the rest of this document. If there is anything you don't understand, be sure to ask your study doctor or nurse.

## What is the purpose of this study?

The purpose of this study is to test the safety of ipatasertib at different doses. "Doses" is defined as the amount of drug you get, We want to find out what effects the drug has on people, if any. There will be around 21-36 people taking part in this study.

# What are the study groups?

There are two parts in this study, a dose escalation part and a dose expansion part. Your doctor will tell you which part you are in.

In the dose escalation part of this study, different people will get different doses of the study drug Ipatasertib. The dose escalation phase of this trial has ended as of **December 22, 2023**.

The first 3 people taking part in this study will get the lowest dose. If the drug does not cause serious side effects, the next group of people in the study will get a higher dose. The study doctor will watch each group carefully as they increase the dose. The doses will continue to increase for every new group until people have serious side effects that require the dose to be lower. Once this dose is found, the dose escalation is stopped. The highest dose with manageable side effects was determined to be of ipatasertib. (22-DEC-2023)

In the dose expansion part of this study, the highest dose with manageable side effects will be of ipatasertib given to 12 more people. This will help study doctors better understand the side effects that may happen with this drug. (22-DEC-2023)


NRG-GY027

- 4 -

Treatment schedule: You will get paclitaxel and carboplatin through a vein in your arm on the first day of each cycle. Each cycle lasts 21 days. This study has 3 cycles.

You will not be able to get additional doses of the study drug. This drug is not approved by the FDA for treatment of your disease.

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.



# What exams, tests, and procedures are involved in this study?

Before you begin the study, your doctor will review the results of your exams, tests, and procedures. This helps your doctor decide if it is safe for you to take part in the study. If you join the study, you will have more exams, tests, and procedures to closely monitor your safety and health. Most of these are included in the usual care you would get even if you were not in a study.

Listed below are tests and procedures needed for research only:

- Collect some of the tissue left over from your previous biopsy or procedure when you
  were diagnosed with cancer and from the surgery you have while on this study.
- Collect some of your blood at two times, before you start the study treatment and when you have surgery on this study.

These samples will be used for research only to identify changes in the tumor and/or blood that may help doctors in the future predict if patients will respond to these study drugs. You and your study doctor will not get the results of this.


NRG-GY027

- 5 -

# What risks can I expect from taking part in this study? General Risks

If you choose to take part in this study, there is a risk that adding the study drug may not be as good as the usual approach alone for your cancer or condition at shrinking or stabilizing your cancer.

You also may have the following discomforts:

- Spend more time in the hospital or doctor's office.
- Be asked sensitive or private questions about things you normally do not discuss.
- May not be able to take part in future studies.

The drugs used in this study could be very harmful to an unborn or newborn baby. There may be some risks that doctors do not yet know about. It is very important that you check with your study doctor about what types of birth control or pregnancy prevention to use during the study and for 28 days after completing your last dose of ipatasertib.

This study will use a sample of your tissue. Generally, your hospital will keep some of your tissue. This tissue may be used to help treat your cancer in the future. Because this study will need to use some of this tissue, there is a small risk that it could be used up.

#### **Genetic Testing Risks**

The genetic test used in this study will test your tumor tissue and blood for genetic changes. Changes found in your normal tissue may be passed down in families. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down.

Since this study is only testing tumor tissue, we will not know if a genetic change in your tumor is also in your normal tissue. If you want to find out if the change is in your normal tissue, then you will need to get other tests done outside of this study.

Genetic tests of normal tissue can reveal information about you and also about your relatives. Your doctor will talk with you about what the tests results may mean for you and your family. He or she also may suggest you talk with a genetics counselor to learn more. You or your insurance plan would have to pay for any genetic tests and visits to a genetic counselor done outside of this study.


#### Side Effect Risks

The drugs used in this study may affect how different parts of your body work such as your liver, kidneys, heart, and blood. The study doctor will test your blood and let you know if changes occur that may affect your health.

There is also a risk that you could have other side effects from the study drugs. Here are important things to know about side effects:

- 1. The study doctors do not know who will or will not have side effects.
- 2. Some side effects may go away soon, some may last a long time, and some may never go
- 3. Some side effects may make it hard for you to have children.
- 4. Some side effects may be mild. Other side effects may be very serious and even result in death.

You can ask your study doctor questions about side effects at any time. Here are important ways to make side effects less of a problem:

- If you notice or feel anything different, tell your study doctor. He or she can check to see if it is a side effect.
- Your study doctor will work with you to treat your side effects.
- Your study doctor may adjust the study drugs to try to reduce side effects.

This study is looking at a combination of the usual drugs used to treat this type of cancer plus a study drug. This different combination of drugs may increase your side effects or may cause new side effects.

#### **Drug Risks**

The tables below show the most common and most serious side effects doctors know about. Keep in mind that there might be other side effects doctors do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

#### Possible Side Effects of Carboplatin and Paclitaxel (Table Version Date: April 28, 2021)

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving Carboplatin and Paclitaxel, more than 20 and up to 100 may have:

- Allergic reaction which may cause rash, low blood pressure, wheezing, shortness of breath, swelling of the face or throat
- Infection, especially when white blood cell count is low
- Bruising, bleeding
- Anemia which may cause tiredness, or may require blood transfusions
- Sores in mouth which may cause difficulty swallowing
- Diarrhea, nausea, vomiting


NRG-GY027

- 7 -

#### COMMON, SOME MAY BE SERIOUS

In 100 people receiving Carboplatin and Paclitaxel, more than 20 and up to 100 may have:

- Muscle weakness
- Numbness, tingling, or pain of the arms, legs, fingers, or toes
- Hair loss

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving Carboplatin and Paclitaxel, from 4 to 20 may have:

- Abnormal heartbeat
- Blood clot which may cause swelling, pain, shortness of breath
- Damage to the lungs which may cause shortness of breath
- Constipation, belly pain
- Changes in taste

#### RARE, AND SERIOUS

In 100 people receiving Carboplatin and Paclitaxel, 3 or fewer may have:

- Heart attack or heart failure which may cause shortness of breath, swelling of ankles, and tiredness
- A tear or a hole in the stomach which may cause belly pain or that may require surgery
- Visual loss
- Difficulty hearing
- Stevens Johnson Syndrome which may cause severe skin rash with blisters and peeling which can involve mouth and other parts of the body

#### Risk Profile for Ipatasertib (CAEPR Version 2.0, September 16, 2021)

#### **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving ipatasertib, more than 20 and up to 100 may have:

- Diarrhea, nausea
- Hyperglycemia

#### OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving ipatasertib, from 4 to 20 may have:

- Anemia which may require blood transfusion
- Pain
- Heartburn, vomiting
- Tiredness
- Loss of appetite
- Changes in taste
- Rash

#### RARE, AND SERIOUS

In 100 people receiving ipatasertib, 3 or fewer may have:

- 8 -


- Sores in the mouth, which may cause difficulty swallowing
- Liver damage which may cause yellowing of the eyes and skin
- Bruising, bleeding
- Damage to the lungs, which may cause shortness of breath

## **Additional Drug Risks**

The study drug could interact with other drugs or certain foods. Your study doctor will give you a drug information wallet card that lists these possible interactions. Share this information with your family members, caregivers, other health care providers, and pharmacists. You will be provided a Patient Drug Interactions Handout.

Rarely, there are problems getting enough supplies of the study drug. If that happens, your doctor will talk with you about your options.

## What are my responsibilities in this study?

If you choose to take part in this study you will need to:

- Keep your study appointments.
- Tell your doctor about:
  - o all medications and supplements you are taking
  - o any side effects
  - o any doctors' visits or hospital stays outside of this study
  - o if you have been or are currently in another research study.
- Write down in your medication diary when you take the study drug at home.
- Carry the provided wallet card at all times and show it to all your healthcare providers

Do not get pregnant or breastfeed while taking part in this study. Tell your study doctor right away if you think that you have become pregnant during the study or within 28 days after your last dose of study drug.

# What are the costs of taking part in this study?

You and/or your insurance plan will need to pay for the costs of medical care you get as part of the study, just as you would if you were getting the usual care for your cancer. This includes:

- The costs of tests, exams, procedures, and drugs that you get during the study to monitor your safety, and prevent and treat side effects.
- The costs of getting the paclitaxel, carboplatin, and ipatasertib ready and giving it to you.
- Your insurance co-pays and deductibles.


NRG-GY027

- 9 -

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it doesn't pay for if you take part in this clinical trial. Also, find out if you need approval from your plan before you can take part in the study.

Ask your doctor, nurse, or study staff for help finding the right person to talk to if you are unsure which costs will be billed to you or your insurance provider.

You and/or your insurance provider will not have to pay for exams, tests, and procedures done for research purposes only or that are covered by the study.

You or your insurance provider will not have to pay for the ipatasertib while you take part in this study.

You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

Taking part in this study may mean that you need to make more visits to the clinic or hospital than if you were getting the usual approach to treat your cancer. You may:

- Have more travel costs.
- Need to take more time off work.
- Have other additional personal costs.

## What happens if I am injured because I took part in this study?

If you are injured as a result of taking part in this study and need medical treatment, please talk with your study doctor right away about your treatment options. The study sponsors will not pay for medical treatment for injury. Your insurance company may not be willing to pay for a study-related injury. Ask them if they will pay. If you do not have insurance, then you would need to pay for these medical costs.

If you feel this injury was caused by medical error on the part of the study doctors or others involved in the study, you have the legal right to seek payment, even though you are in a study. Agreeing to take part in this study does not mean you give up these rights.

# Who will see my medical information?

Your privacy is very important to us. The study doctors will make every effort to protect it. The study doctors have a privacy permit to help protect your records if there is a court case. However, some of your medical information may be given out if required by law. If this should happen, the study doctors will do their best to make sure that any information that goes out to others will not identify who you are.

Some of your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the study sponsor in a central research database. However, your name and contact information will not be put in the database. If information

- 10 -


from this study is published or presented at scientific meetings, your name and other personal information will not be used.

There are organizations that may look at or receive copies of some of the information in your study records. Your health information in the research database also may be shared with these organizations. They must keep your information private, unless required by law to give it to another group.

Some of these organizations are:

- The study sponsor, National Cancer Institute- Cancer Therapy Evaluation Program (NCI-CTEP) and any company supporting the study now or in the future. This would include any organization helping the company with the study.
- The NCI Central IRB, which is a group of people who review the research with the goal of protecting the people who take part in the study.
- The FDA and the groups it works with to review research.
- The NCI and the groups it works with to review research.
- The NCI's National Clinical Trials Network and the groups it works with to conduct research, including NRG Oncology and the Imaging and Radiation Oncology Core (IROC).
- The NRG Oncology Biospecimen Bank-Columbus (Biobank) and laboratories designated by NRG Oncology to perform testing as part of the study.

In addition to storing data in the study database, data from studies that are publicly funded may also be shared broadly for future research with protections for your privacy. The goal of this data sharing is to make more research possible that may improve people's health. Your study records may be stored and shared for future use in public databases. However, your name and other personal information will not be used.

Some types of future research may include looking at your information and information from other patients to see who had side effects across many studies or comparing new study data with older study data. However, right now we don't know what research may be done in the future using your information. This means that:

- You will not be asked if you agree to take part in the specific future research studies using your health information.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your information.

There are laws that protect your genetic information. However, there is a risk that someone could get access to your genetic information and identify you by name. In some cases, employers could use your genetic information to decide whether to hire or fire you. The study doctors believe the risk of this happening is very small. However, the risk may increase in the future as people find new ways of tracing information. For more information about the laws that protect you, ask your study doctor.

- 11 -


## Where can I get more information?

You may visit the NCI web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns you have about this study or to report side effects or injuries. Contact the study doctor (\*insert name of study doctor[s]\*) at (\*insert telephone number, and email address if appropriate\*).

For questions about your rights while in this study, call the (\*insert name of organization or center\*) Institutional Review Board at (\*insert telephone number\*).

## Optional studies that you can choose to take part in

# Optional sample collections for known laboratory studies and/or storage for possible future studies

Researchers are trying to learn more about cancer and other health problems using blood and tissue samples from people who take part in clinical trials. By studying these samples, researchers hope to find new ways to prevent, detect, treat, or cure diseases.

Some of these studies may be about how genes affect health and disease. Other studies may look at how genes affect a person's response to treatment. Genes carry information about traits that are found in you and your family. Examples of traits are the color of your eyes, having curly or straight hair, and certain health conditions that are passed down in families. Some of the studies may lead to new products, such as drugs or tests for diseases.

#### **Known future studies**

If you choose to take part in this optional study, researchers will collect some of your blood for research on the diversity of your immune cells. Your study doctor will collect some of your blood at two times during the study – Before you start study treatment and when you have the surgery on this trial. If you agree, your study doctor may also submit an additional sample of your tumor tissue, as well of some of your normal tissue, that may have been collected during your previous biopsy or procedure when you were diagnosed with cancer. These tissue samples will be used for research to identify changes in the tumor and/or blood that may help doctors in the future predict if patients will respond to these study drugs.

#### Unknown future studies

- 12 -


If you choose to take part in this optional study, any tissue and blood remaining after the research described will be stored. Storing samples for future studies is called "biobanking." The biobank is being run by NRG Oncology and is supported by the NCI. This is a publicly funded study. Samples from publicly funded studies are required to be shared as broadly as possible. However, we will protect your privacy. The goal of this is to make more research possible that may improve people's health.

The biobank is a public research resource. It has controlled access. This means that researchers who want to get samples and data from it must submit a specific research request. The request identifies who they are and what their planned research project is. Before getting the samples and data, the researchers must agree to keep the data private, only use it for their planned research project, and never use it to try to identify you.

Right now, we don't know what research may be done in the future using your tissue and blood samples. This means that:

- You will not be asked if you agree to take part in the future research studies.
- You and your study doctor will not be told when or what type of research will be done.
- You will not get reports or other information about any research that is done using your samples.

Unknown future research studies may include sequencing of all or part of your DNA. This is called genomic sequencing. Sequencing allows researchers to identify your genetic code. Changes in your genetic code may just be in your tumor tissue. These are called somatic changes. Changes may also be in your normal tissue and passed down through your family. For example, these genetic changes may be passed down to your children in the same way that eye and hair color are passed down. These are called germline changes. If only tumor tissue is sequenced, we will not know if a genetic change in your tumor is also in your normal tissue. This is why sometimes both normal tissue and tumor tissue are sequenced. This helps researchers understand if a genetic change happened only in your cancer tissue, or in your normal tissue as well.

#### What is involved in this optional sample collection?

If you agree to take part, here is what will happen next:

- 1. About one teaspoon of blood will be collected from a vein in your arm at two different times Before you start study treatment and when you have the surgery on this trial.
- 2. Any tissue and blood remaining after the research described will be stored in the biobank. There is no limit on the length of time we will keep your samples and research information. The samples will be kept until they are used for research or destroyed.
- 3. Researchers can only get samples from the biobank after their research has been approved by experts. Researchers will not be given your name or contact information.
- 4. Some of your genetic and health information may be placed in central databases for researchers to use. The databases will not include your name or contact information.

- 13 -


#### What are the risks in this optional sample collection?

- The most common risks related to drawing blood from your arm are brief pain and maybe a bruise.
- Generally, hospitals will keep some of your tissue. This tissue may be used to help treat your cancer in the future. There is a small risk that when this tissue sample is submitted to the biobank for this optional sample collection, your tissue could be used up.
- Your medical and genetic information is unique to you. There is a risk that someone
  outside of the research study could get access to your study records or trace information
  in a database back to you. They could use that information in a way that could harm you.
  Researchers believe the chance that someone could access and misuse your information is
  very small. However, the risk may increase in the future as people find new ways of
  tracing information.
- In some cases, this information could be used to make it harder for you to get or keep a job and get or keep health insurance. There are laws against the misuse of genetic information, but they may not give full protection. For more information about the laws that protect you, ask your study doctor or visit: https://www.genome.gov/10002328/

## How will information about me be kept private?

Your privacy is very important to the study researchers and biobank. They will make every effort to protect it. Here are just a few of the steps they will take:

- 1. They will remove identifiers, such as your initials, from your sample and information. They will replace them with a code number. There will be a master list linking the code numbers to names, but they will keep it separate from the samples and information.
- 2. Researchers who study your sample and information will not know who you are. They also must agree that they will not try to find out who you are.
- 3. Your personal information will not be given to anyone unless it is required by law.
- 4. If research results are published, your name and other personal information will not be used.

#### What are the benefits to taking part in this optional sample collection?

You will not benefit from taking part.

The researchers, using the samples from you and others, might make discoveries that could help people in the future.

## Are there any costs or payments to this optional sample collection?

There are no costs to you or your insurance. You will not be paid for taking part in this study. The research may lead to new tests, drugs, or other products for sale. If it does, you will not get any payment.

## What if I change my mind about this optional sample collection?

- 14 -


If you decide you no longer want your samples to be used, you can call the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*), who will let the biobank know. Then, any sample that remains in the biobank will be destroyed or returned to your study doctor. This will not apply to any samples or related health information that have already been given to or used by researchers.

## What if I have questions about this optional sample collection?

If you have questions about the use of your samples for research, contact the study doctor, (\*insert name of study doctor for main trial\*), at (\*insert telephone number of study doctor for main trial\*).

Please circle your answer below to show if you would or would not like to take part in each optional study.

#### Samples for known future studies:

I agree that my samples and related health information may be used for the laboratory study described above.

YES NO

## Samples for unknown future studies:

I agree that my samples and related health information may be kept in a biobank for use in future health research.

YES NO

#### **Contact for Future Research**

I agree that my study doctor, or someone on the study team, may contact me or my doctor to see if I wish to participate in other research in the future.

YES NO

This is the end of the section about optional studies.


## My signature agreeing to take part in the study

I have read this consent form or had it read to me. I have discussed it with the study doctor and my questions have been answered. I will be given a signed and dated copy of this form. I agree to take part in the main study. I also agree to take part in any additional studies where I circled "yes".

| Participant's Printed Nan | ne |
|---------------------------|-------------------------------------------|
| Participant's signature _ | |
| Date of signature | |
| Signature of person(s) o | onducting the informed consent discussion |
| Printed Name | |
| Signature | |
| Date of signature | |
